CLINICAL TRIAL: NCT02825810
Title: Effectiveness of a Physical Therapy Program for Improving Cervical Motor Control in Long-term Breast Cancer Survivors
Brief Title: Cervical Motor Control in Long-term Breast Cancer Survivors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding issues, poor prevalence of low cervical motor control
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Irene Cantarero Villanueva, PhD, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UGR0116
Record Dates: First submitted 2016-07-04; First posted 2016-07-07 (Estimated); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; long-term survival; motor control; cervical pain
MeSH Terms: conditions — Breast Neoplasms; Neck Pain

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Cervical motor control group (Experimental)
  Interventions: Behavioral: Cervical motor control
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Cervical motor control — Intervention will consist in a tailored exercise training following a previous published motor control protocol
  Arms: Cervical motor control group

SUMMARY:
The aim of this study will be to determine the effectiveness of a physical therapy program which is based on cervical motor control exercises in long-term breast cancer survivors in order to improve their motor control and its possible impact on pain, mood state and quality of life.

DETAILED DESCRIPTION:
Background: Breast cancer is becoming a common disease; however survival rates have improved throughout the last years. As a result, this also means that breast cancer survivors suffer side effects concerning the disease itself and treatments, as it is the case of certain kinds of pain. It is known that 80% of breast cancer survivors suffer this even 5 years after the completion of treatment and this impairment can be associated with a high tendency towards depression, cardiorespiratory deconditioning and even altered cervical control motor.

Aim: To determine the effectiveness of a physical therapy program based on cervical motor control training in order to improve motor control, mood state and quality of life.

Methods: Fifty-two long-term breast cancer survivors will be allocated to experimental group (n=26) or control group (n=26). The experimental group will receive a nine-week tailored exercise training focused on cervical motor control.

Discussion: There is a lack of knowledge about effective interventions when it comes to deal with altered motor control pattern of cervical area in long-term breast cancer survivors. Therefore, it is necessary to study the impact of this novel approach to improve quality of life in this population.

ELIGIBILITY:
Inclusion Criteria:

* To be over 18 years old
* Have passed a period equal o more 5 years since breast cancer diagnosis
* Have diagnosis of stage I, II or IIIA breast cancer
* Have signed informed consent
* Have medical clearance for participation
* Inability to get level 2 in the craniocervical flexion test

Exclusion Criteria:

* Have diagnosis of arthritis or fibromyalgia
* Have cancer recurrence
* Have been operated through previous surgery of cervical column
* To be taking any treatment for pain or altered motor control during last 12 months

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10; Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index (NDI) | Participants will be followed over 9 weeks
  It is self-administered questionnaire to test neck pain interference in daily activities. It contains 10 items

SECONDARY OUTCOMES:
Craniocervical Flexion Test (CCFT) | Participants will be followed over 9 weeks
  It is used to assess deficit of cervical motor pattern
Algometry | Participants will be followed over 9 weeks
  Pressure pain thresholds (PPTs) will be assessed using an electronic algometer (Somedic AB, Farsta, Sweden)
Visual Analogue Scale (VAS) | Participants will be followed over 9 weeks
  It is used to assess subjective pain. It contains scores in the range of 0 to 10 (0 = 'no pain'; 10 = 'worst imaginable pain'). Participants will have to mark the level of pain that they feel in that moment for neck-shoulders areas
Scale for Mood Assessment | Participants will be followed over 9 weeks
  It is used to assess 4 moods: anxiety, anger-hostility, sadness-depression, and happiness. It contains 16 items
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) version 3.0 | Participants will be followed over 9 weeks
  It is used to asses quality of life. It contains 30 items with both multi-item scales and single-item measures
European Organization for Research and Treatment of Cancer Breast Cancer-Specific Quality of Life Questionnaire (EORTC QLQ-BR23) | Participants will be followed over 9 weeks
  It is a breast cancer module of EORTC QLQ-C30. This module contains 23 items assessing disease symptoms, side effects of treatment, body image, sexual functioning, and future perspective
Minnesota Leisure Time Physical Activity Questionnaire (MLTPAQ) | Participants will be followed over 9 weeks
  It is used to calculate energy expenditure for leisure time physical activity
International Fitness Scale (IFIS) | Participants will be followed over 9 weeks
  It is used to assess perceived patients' overall fitness, cardio-respiratory fitness, muscular fitness, speed-agility and flexibility

CONTACTS AND LOCATIONS:
Overall Officials: Irene Cantarero-Villanueva, PhD, Principal Investigator — Physical Therapy Deparment, Faculty of Health Sciences, University of Granada
Locations (1):
- University of Granada, Granada, Spain